CLINICAL TRIAL: NCT05154292
Title: A Serious Game for Psychological Assessment and Intervention in Adolescents With Emotional Regulation Problems
Brief Title: SAEM: A Serious Game for Emotional Regulation Problems in Adolescents
Acronym: SAEMGame
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universidad de Almeria (Other)
Collaborators: Universitat Jaume I (Other); Fundación Pública Andaluza para la Investigación Biomédica Andalucía Oriental (Other)
Responsible Party: Principal Investigator, Juan Miguel Flujas, PhD, Universidad de Almeria
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: UALPsy002
Record Dates: First submitted 2021-11-29; First posted 2021-12-13 (Actual); Last update posted 2021-12-13 (Actual); Status verified 2021-11

CONDITIONS: Adolescents
Keywords: Emotion Regulation; Adolescents; Serious Game; Anxiety; Behavior problems
MeSH Terms: conditions — Emotional Regulation; Anxiety Disorders; Mental Disorders

STUDY DESIGN:
Intervention Model Description: Clinical Trial
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- eHealth Emotion Regulation Skills (Experimental): The intervention aims to develop competencies for emotional regulation through exposure and acceptance strategies for coping with circumstances that produce stress or emotional discomfort. The application has a series of mini-games that the user will overcome throughout a narrative, with different challenges and rewards
  Interventions: Behavioral: Serious Game: Emotional Health Island (SAEM)
- Waiting List (No Intervention): He or she will not be exposed to the intervention but will remain on the waiting list and will complete the pre and post-measures.

INTERVENTIONS:
Behavioral: Serious Game: Emotional Health Island (SAEM) — This intervention aims to aim to develop competencies for emotional regulation through exposure and acceptance strategies. This intervention is applied through a serious game developed for this purpose. the adolescent will complete a series of missions aimed at developing skills related to psychological flexibility, namely, greater psychological acceptance, mindfulness in the present moment, and committed actions in the direction of personal values. This serious game is guided by a therapist.
  Other Names: Isla de SAEM (Salud Emocional) (ES)
  Arms: eHealth Emotion Regulation Skills

SUMMARY:
This study aims to assess the effects of an intervention to improve emotional regulation skills in adolescents with affective (anxiety and/or depression) and behavioral problems.

DETAILED DESCRIPTION:
Emotional regulation skills and strategies are a protective factor against various problems and psychopathologies. The development and maintenance of affective symptoms are usually very harmful to the adolescent and for his/her family and social environment and can lead to other more serious psychological problems (depression, anxiety, adaptive disorders, etc.) or problems of socio-educational maladjustment.

This study aims to improve the emotional regulation of adolescents who present affective symptoms related to anxiety, depression, or behavioral problems, such as difficulties in their interpersonal relationships, impulsivity, anxiety, anger attacks, low tolerance to frustration, apathy, or sadness. The intervention program, applied through a video game, is an intervention protocol for emotional well-being that has been tested and validated in an adolescent population with emotional and behavioral problems.

ELIGIBILITY:
Inclusion Criteria:

* Between 12 and 16 years old
* Show affective symptoms associated with depression and anxiety or behavior problems
* Show willingness to participate in the research study
* Understand written and spoken Spanish
* Show stability in treatment dosage, if taking medication.

Exclusion Criteria:

* Exhibit incapacitating neurological and/or intellectual impairment
* Have a diagnosis of severe mental disorder
* Substance abuse addiction or dependence

Ages: 12 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 120 (Estimated)
Dates: Start 2022-01-01 (Estimated); Primary Completion 2022-07-30 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
The Difficulties in Emotional Regulation Scale (DERS; Hervás & Jódar, 2008) | Change from baseline at immediately after the intervention, and at 3 months
  Consists of 28 items that make up 6 dimensions of emotional dysregulation: attention, acceptance, impulsivity, clarity, goals and strategies. The reliability index is between .87 and .93.
Revised Child Anxiety and Depression Scale (RCADS-30; Pineda et al., 2018) | Change from baseline at immediately after the intervention, and at 3 months
  it is a 30-item scale to assess the presence of symptoms associated or compatible with depression and anxiety in children and adolescents. Internal consistency between .78 and .93.

SECONDARY OUTCOMES:
Avoidance and Fusion Questionnaire for Young People (AFQ-Y; Valdivia-Salas, Martín-Albo, Zaldívar, Lombas, & Jiménez, 2016) | Change from baseline at immediately after the intervention, and at 3 months
  that assesses the level of avoidance and cognitive fusion present when faced with distressing situations. This scale presents a Cronbach's alpha between .76 and 87.
. Willingness and Action Scale for Children and Adolescents (WAM; Cobos, Flujas-Contreras, & Gomez, 2020) | Change from baseline at immediately after the intervention, and at 3 months
  ) to assess levels of acceptance and behavioral activation (action) in the direction of valued life areas. This scale shows an internal consistency between .76 and .81.
Mood and coping | Change from baseline at immediately after the intervention, and at 3 months
  At the start and close of the App, a series of questions will appear that measure mood of the users by means of a visual face scale (5-point Likert) and a coping question by means of a 5-point Likert scale.

CONTACTS AND LOCATIONS:
Overall Officials: Inmaculada Gómez Becerra, Prof PhD, Principal Investigator — Universidad de Almeria
Locations (3):
- Spain (3):
  - Torrecardenas Hospital, Almería, Andalusia
  - University of Almería, Almería, Andalusia
  - University Jaume I, Castellon, Castellón

IPD SHARING:
Plan to Share IPD: Yes
The data will be published in a data repository and in the publications that are necessary. The data related to the responses will be published in the self-reported evaluation systems, mainly, pre, post and follow-up that have an impact on the evaluation of the effectiveness of the treatment.
Supporting Information: Study Protocol, ICF
Time Frame: At the end of the RCT. For a period of 1 year.
Access Criteria: Open access in data repository or under request to authors.